CLINICAL TRIAL: NCT04292093
Title: Studio di Efficacia di Percorsi di Riabilitazione Neuropsicologica Tramite Piattaforma Lumosity: Evidenze Comportamentali e Neurofisiologiche in Pazienti Con Epilessia Non Sintomatica in età Pediatrica
Brief Title: Efficacy Study of a Neuropsychological Rehabilitation Intervention for Children With Non-symptomatic Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 769
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Children; Rehabilitation; Executive Functions
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home rehabilitation training (Experimental): Home rehabilitation training
  Interventions: Behavioral: Home rehabilitation training
- Home control activity (Active Comparator): Home control activity
  Interventions: Behavioral: Home control activity

INTERVENTIONS:
Behavioral: Home rehabilitation training — The rehabilitation training will be provided via Lumosity platform. Participants will be asked to play computer video-games aimed at strengthening specific sub-functions pertaining to the macro area of executive functions for 30 minutes a day, 5 days a week, for a total of 8 weeks. Specifically, 20 games out of a total of 64 available games provided by the platform have been selected. The selected games are aimed at training 4 cognitive skills: memory, attention, cognitive flexibility and problem solving. In particular, 5 different games were chosen for each cognitive ability.
  Arms: Home rehabilitation training
Behavioral: Home control activity — The control group will watch a series of animated / TV shows suitable for the sample age, again for 30 minutes a day, 5 days a week, for 8 weeks. The videos will be provided by the experimenter and participants will watch them on their personal computer. At the end of each videos, participants will answer a series of multiple-choice questions aimed at evaluating the attention deployed to the content of the videos.
  Arms: Home control activity

SUMMARY:
Patients with non-symptomatic epilepsy, even in the presence of a normative cognitive functioning, present different levels of neuropsychological weaknesses, especially in executive functions and social competences. Such difficulties can significantly influence academic achievement and social inclusion. To date, there is limited evidence on small samples that training focusing on executive functions, also through tele-rehabilitation methods, may be effective in limiting these difficulties. Therefore, the purpose of this research project is to evaluate the effectiveness of a training of the executive functions (administered via the Lumosity platform) in patients with non-symptomatic focal and generalized epilepsy. A cognitive and behavioral assessment will be performed before and after the treatment to evaluate its efficacy. Moreover, a predefined neurophysiological marker will be recorded before and after treatment to detect changes in cortical activity which may reflect expected treatment effects.

DETAILED DESCRIPTION:
First, all eligible patients will be screened for inclusion and exclusion and will be assigned to the experimental group and the control group. The experimental group will participate in a remote rehabilitation program via Lumosity platform, providing video-games aimed at strengthening specific cognitive functions for 30 minutes a day, 5 days a week, for a total of 8 weeks. The control group will watch a series of animated / TV shows, again for 30 minutes a day, 5 days a week, for 8 weeks. Once a week the patient (or his family) will be contacted by the researcher to check the progress of the treatment. All patients will be evaluated within a week before the start of treatment and after the end of treatment with a standardized neuropsychological assessment battery (NEPSY-II) designed to evaluate the effects of the treatment. Patients (or their parents according to participants' age) will also compile a questionnaire to assess behavioral problems (CBCL); a questionnaire for the assessment of cognitive functions in an ecological context (BRIEF-2); a quality of life questionnaire (TACQOL) and ad-hoc treatment appreciation questionnaire. In addition to the cognitive-behavioral assessment, specific parameters of cortical activity will be recorded (via EEG), in order to evaluate any changes in predefined neurophysiological markers able to reflect the effects of the treatment. Evidence gathered from the literature reports that the relationship between theta and beta waves (the so-called theta/beta ratio) may be considered an index of a behavioral adaptation deficit in populations with poor executive control. Therefore, this index appears to be the ideal candidate to detect changes in cortical activity which may underlay behavioral effects of home rehabilitation treatment. Thus, resting-state cortical activity will be recorded before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-symptomatic epilepsy;
* Absence of intellectual disability (total IQ> 70);
* Absence of significant visual, auditory or motor impairments that may prevent the use of the computerized training;
* Basic ability to use PC.

Exclusion Criteria:

* Presence of psychiatric comorbidity and / or behavioral disturbances that may hamper the participation to training sessions;
* Diagnosis of photosensitive epilepsy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
NEPSY-II Neuropsychological Battery | baseline
  Assessment of executive functions, language, memory and visuo-spatial skills
  Subscales (all subscales range from 1 to 19 scalar scores):
  * Design fluency, raw score 0/70
  * Auditory attention, 0/30 and Response Set 0/36
  * Inhibition (denomination 0/80 - 0/360') (inhibition 0/80 - 480') (switching 0/80 - 480') REVERSE (higher raw scores indicate worse perfomance)
  * Animal sorting, 0/12
  * Word generation, 0/75
  * Memory for faces, 0/32
  * Word list interference (repetition 0/20; recall 0/40)
  * Imitating hand position, (0/24)
  * Visuo-motor precision (0/307; 0/360') REVERSE (higher raw scores indicate worse perfomance)
  * Manual motor sequences, 0/60
  * Affect recognition, 0/35
  * Design copying (general 0/21; motor 0/42; global 0/42; local 0/36; total specific 0/120)
  * Picture puzzles, 0/20
  * Geometric puzzles, 0/40
Wechsler Intelligence Scale for Children Fourth Edition (WISC-IV) | baseline
  Assessment of general intellectual ability. Indexes (higher T scores indicate better perfomance for all indexes)
  * Verbal Comprehension Index (40/160)
  * Fluid Reasoning Index (40/160)
  * Working Memory Index (40/160)
  * Processing Speed Index (40/160)
  * Full Scale IQ (40/160)
NEPSY-II Neuropsychological Battery (change) | within 1 week after intervention
  Assessment of executive functions, language, memory and visuo-spatial skills
NEPSY-II Neuropsychological Battery (change) | 3 month after intervention
  Assessment of executive functions, language, memory and visuo-spatial skills

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) (parent compiled for 6-18 years old participants) | baseline
  Questionnaire for the assessment of emotional and behavioural problems.
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self Report (CBCL self-report version for 11-18 years old participants) | baseline
  Questionnaire for the assessment of emotional and behavioural problems.
  YSR 11-18 is direcly compiled by adolescents aged 11-18 years. It provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
The Children's Quality of Life (TACQOL) | baseline
  Questionnaire for the assessment of health-related quality of life.
  Scales (higher raw scores indicate higher quality of life)
  * Body (physical functioning) 0/32
  * Motor functioning 0/32
  * Autonomy 0/32
  * Social functioning 0/32
  * Cognition 0/32
  * Emotions (positive) 0/16
  * Emotions (negative) 0/16
Behavior Rating Inventory of Executive Function (BRIEF-2) (parent compiled for 5-10 years old participants; self-report version for 11-18 years old participants) | baseline
  Questionnaire for the assessesment of executive function and self-regulation competence.
  The BRIEF (parent version) questionnaire is aimed at assessing executive functioning at home and school and contains 63 items. Raw scores of the global scale range from 63 to 189; T scores (M = 50, SD = 10). The self-report version contains 55 items. Raw scores of the global scale range from 55 to 165; T scores (M = 50, SD = 10). Higher scores mean a worse outcome.
  Subscale and Indexes
  * Inhibit
  * Shift
  * Self-Monitor
  * Emotional Control
  * Initiate
  * Working Memory
  * Plan/Organize
  * Behavioral regulation Index
  * Emotion regulation Index
  * Cognitive regulation Index
  * Global Executive Index
Theta/beta ratio | baseline
  Low theta/beta ratio is a cortical activity considered an index of poor attentional resources. Its recording will be conducted with a 32-channels EEG system at rest (4 minutes: 2 min eyes open and 2 min eyes closed).
Child Behavior Checklist CBCL (change) | within 1 week after intervention
  Questionnaire for the assessment of emotional and behavioural problems
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self Report (CBCL self-report version for 11-18 years old participants) | within 1 week after intervention
  Questionnaire for the assessment of emotional and behavioural problems.
  YSR 11-18 is direcly compiled by adolescents aged 11-18 years. It provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
The Children's Quality of Life TACQOL (change) | within 1 week after intervention
  Questionnaire for the assessment of health-related quality of life. Scales (higher raw scores indicate higher quality of life)
  * Body (physical functioning) 0/32
  * Motor functioning 0/32
  * Autonomy 0/32
  * Social functioning 0/32
  * Cognition 0/32
  * Emotions (positive) 0/16
  * Emotions (negative) 0/16
Behavior Rating Inventory of Executive Function (BRIEF-2) (change) | within 1 week after intervention
  Questionnaire for the assessesment of executive function and self-regulation competence.
  The BRIEF (parent version) questionnaire is aimed at assessing executive functioning at home and school and contains 63 items. Raw scores of the global scale range from 63 to 189; T scores (M = 50, SD = 10). The self-report version contains 55 items. Raw scores of the global scale range from 55 to 165; T scores (M = 50, SD = 10). Higher scores mean a worse outcome.
  Subscale and Indexes
  * Inhibit
  * Shift
  * Self-Monitor
  * Emotional Control
  * Initiate
  * Working Memory
  * Plan/Organize
  * Behavioral regulation Index
  * Emotion regulation Index
  * Cognitive regulation Index
  * Global Executive Index
Theta/beta ratio (change) | within 1 week after intervention
  Low theta/beta ratio is a cortical activity considered an index of poor attentional resources. Its recording will be conducted with a 32-channels EEG system at rest (4 minutes: 2 min eyes open and 2 min eyes closed).
Ad-hoc compliance to treatment questionnaire | within 1 week after intervention
  A 5 items of a 5-point Likert questionnaire created ad-hoc for the assessment of the compliance to the treatment.
  Higher scores indicare better compliance (except for item 4)
Child Behavior Checklist CBCL (change) | 3 months after intervention
  Questionnaire for the assessment of emotional and behavioural problems
  The CBCL 6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 DSM-oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
Youth Self Report (CBCL self-report version for 11-18 years old participants) | 3 month after intervention
  Questionnaire for the assessment of emotional and behavioural problems.
  YSR 11-18 is direcly compiled by adolescents aged 11-18 years. It provides a total score, an internalizing score and an externalizing score, together with eight empirically based syndromes and DSM-oriented scales. It contains 112 items. Raw scores of the Total Problems Scale range from 0 to 224. T scores (M = 50, SD = 10) are used to interpret the level of behavioral functioning. Higher scores mean a worse outcome.
The Children's Quality of Life TACQOL (change) | 3 months after intervention
  Questionnaire for the assessment of health-related quality of life.
  Scales (higher raw scores indicate higher quality of life)
  * Body (physical functioning) 0/32
  * Motor functioning 0/32
  * Autonomy 0/32
  * Social functioning 0/32
  * Cognition 0/32
  * Emotions (positive) 0/16
  * Emotions (negative) 0/16
Behavior Rating Inventory of Executive Function (BRIEF-2) (change) | 3 month after intervention
  Questionnaire for the assessesment of executive function and self-regulation competence.
  The BRIEF (parent version) questionnaire is aimed at assessing executive functioning at home and school and contains 63 items. Raw scores of the global scale range from 63 to 189; T scores (M = 50, SD = 10). The self-report version contains 55 items. Raw scores of the global scale range from 55 to 165; T scores (M = 50, SD = 10). Higher scores mean a worse outcome.
  Subscale and Indexes
  * Inhibit
  * Shift
  * Self-Monitor
  * Emotional Control
  * Initiate
  * Working Memory
  * Plan/Organize
  * Behavioral regulation Index
  * Emotion regulation Index
  * Cognitive regulation Index
  * Global Executive Index

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Bardoni, MD, PhD, Principal Investigator — Scientific Institute, IRCCS E. Medea